CLINICAL TRIAL: NCT06243978
Title: Effectiveness of a Digital Health Application for Primary Hypertension (Liebria): Randomized Controlled Trial
Brief Title: Effectiveness of a Digital Health Application for Primary Hypertension (Liebria)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: liebria RCT 2024
Record Dates: First submitted 2024-01-17; First posted 2024-02-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liebria (Experimental): Participants allocated to the intervention group will receive access to liebria in addition to treatment as usual (TAU).
  reviga is a digital health application designed for individuals with hypertension, accessible through a web browser. The application focuses on evidence-based psychological and psychotherapeutic methods combined with psychoeducation and health behavior change. Topics addressed by liebria include clarifying and strengthening motivation, training the parasympathetic nervous system, recognizing and overcoming obstacles, strengthening impulse control, development of an individualized day plan, and relapse prevention.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivating text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 360 days.
  Interventions: Behavioral: liebria
- brochure on hypertension (Other): Participants allocated to the control group will receive a brochure from the Deutsche Hochdruckliga (German Hypertension League) in addition to TAU.
  Interventions: Other: information brochure on hypertension

INTERVENTIONS:
Behavioral: liebria — Participants will receive access to the digital health intervention liebria in addition to TAU
  Arms: liebria
Other: information brochure on hypertension — Participants will receive an information brochure on hypertension
  Arms: brochure on hypertension

SUMMARY:
This clinical trial with 328 patients with primary hypertension aims to investigate the effectiveness of the self-guided digital application liebria for patients with primary hypertension.

DETAILED DESCRIPTION:
This clinical trial with 328 patients with primary hypertension aims to investigate the effectiveness of the self-guided digital application liebria for patients with primary hypertension. Inclusion criteria are: age ≥ 18; presence of primary hypertension (confirmed by medical certificate or equivalent); unmedicated or with existing antihypertensive drug therapy (with stable dose in the past 6 weeks prior to study enrolment); last reported office-based systolic blood pressure (SBP) ≥ 140 mmHg followed by home-based SBP ≥ 135 mmHg; consent to participate. Exclusion criteria are: home-based SBP > 180 mmHg; > triple combination of antihypertensive medication; history of secondary hypertension (e.g., thyroid disease, kidney disease); pregnancy.

Patients will be randomized and allocated in a 1:1 ratio to either an intervention group, in which they will receive access to liebria in addition to treatment as usual (TAU, n = 164), or to a control group, in which they will receive a relevant brochure from the Deutsche Hochdruckliga (German Hypertension League) in addition to TAU (n = 164). TAU is defined as any therapy prescribed or recommended by the GP or specialists (e. g. cardiologist).

The primary endpoint will be home-based SBP, with 6 months post-allocation being the primary time point for assessment of effectiveness. Three months post-allocation will be used as an additional endpoint. Secondary endpoints will be patient activation, social and work-related functioning, medication adherence, home-based diastolic blood pressure (DBP), and pulse pressure.

Analysis of effectiveness of the intervention will be performed by ANCOVA of the primary endpoint and all secondary endpoints, in which the posttreatment scores will be compared between treatment groups (intervention group vs. control group), using the baseline scores of the respective outcome as a covariate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Presence of primary hypertension, confirmed by submission of a medical certificate or equivalent (e.g., informal letter signed by primary care physician); relevant ICD-10-GM diagnoses:

  * I10.00 (Benign essential hypertension: Without indication of hypertensive crisis)
  * I10.90 (Essential hypertension, unspecified: Without indication of hypertensive crisis)
* Unmedicated or with existing antihypertensive drug therapy (with stable dose in the past 6 weeks prior to study enrolment)
* Last reported office-based systolic blood pressure (SBP) ≥ 140 mmHg followed by home-based SBP ≥ 135 mmHg
* Consent to participate

Exclusion Criteria:

* Home-based SBP > 180 mmHg
* > Triple combination of antihypertensive medication
* History of secondary hypertension (e.g., thyroid disease, kidney disease)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
SBP (in mmHg) | 6 months
  The primary endpoint is SBP collected via home-based blood pressure measurement (HBPM) using a validated semi-automatic arm cuff device. HBPM will be performed according to the recommendations of the European Society of Hypertension.

SECONDARY OUTCOMES:
Patient activation | 6 months
  Patient Activation Measure (PAM-13). Total score ranging from 0-100; higher scores mean higher activation (better outcome).
Social and work-related functioning | 6 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher impairment (worse outcome).
Adherence to medication | 6 months
  Rief Adherence Index (RAI). Total score ranging from 4-20; higher scores mean higher non-adherence (worse outcome).
DBP (in mmHg) | 6 months
  DBP is collected via home-based blood pressure measurement (HBPM) using a validated semi-automatic arm cuff device. HBPM will be performed according to the recommendations of the European Society of Hypertension.
Pulse pressure (in mmHg) | 6 months
  Pulse pressure (PP) is collected via home-based blood pressure measurement (HBPM) using a validated semi-automatic arm cuff device. HBPM will be performed according to the recommendations of the European Society of Hypertension.

OTHER OUTCOMES:
Body Mass Index | 6 months, 3 months
  weight in kilograms and height in meters will be assessed and combined to report BMI in kg/m^2
concomitant antihypertensive medication | 6 months, 3 months
  number and dosage of concomitant antihypertensive medications (agents in section C of the Anatomical Therapeutic Chemical Classification System)
24-hour average SBP (in mmHg) | 6 months, 3 months
  A 24-hour ambulatory blood pressure measurement (ABPM) will be performed according to recommendations of the International Society of Cardiology: ABPM will be conducted using an FDA-cleared, CE-labeled wireless, non-invasive chest-patch sensor for 24-hour, with measurements four times an hour over 24-hours, resulting in a total of 96 possible measurements.
24-hour average DBP (in mmHg) | 6 months, 3 months
  A 24-hour ambulatory blood pressure measurement (ABPM) will be performed according to recommendations of the International Society of Cardiology: ABPM will be conducted using an FDA-cleared, CE-labeled wireless, non-invasive chest-patch sensor for 24-hour, with measurements four times an hour over 24-hours, resulting in a total of 96 possible measurements.
24-hour average PP (in mmHg) | 6 months, 3 months
  A 24-hour ambulatory blood pressure measurement (ABPM) will be performed according to recommendations of the International Society of Cardiology: ABPM will be conducted using an FDA-cleared, CE-labeled wireless, non-invasive chest-patch sensor for 24-hour, with measurements four times an hour over 24-hours, resulting in a total of 96 possible measurements.
Daytime average SBP (in mmHg) | 6 months, 3 months
  Daytime average SBP will be defined as the average of those ABPM measurements collected between 10:00 and 20:00, in agreement with the International Database of ABP in relation to Cardiovascular Outcome (IDACO) criteria for Europeans.
Nighttime average SBP (in mmHg) | 6 months, 3 months
  Nighttime average SBP will be defined as the average of those ABPM measurements collected between 0:00 and 06:00, in agreement with the IDACO criteria for Europeans
SBP (in mmHg) | 3 months
  The primary endpoint is SBP collected via home-based blood pressure measurement (HBPM) using a validated semi-automatic arm cuff device. HBPM will be performed according to the recommendations of the European Society of Hypertension.
Patient activation | 3 months
  Patient Activation Measure (PAM-13). Total score ranging from 0-100; higher scores mean higher activation (better outcome).
Social and work-related functioning | 3 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher impairment (worse outcome).
Adherence to medication | 3 months
  Rief Adherence Index (RAI). Total score ranging from 4-20; higher scores mean higher non-adherence (worse outcome).
DBP (in mmHg) | 3 months
  DBP is collected via home-based blood pressure measurement (HBPM) using a validated semi-automatic arm cuff device. HBPM will be performed according to the recommendations of the European Society of Hypertension.
Pulse pressure (in mmHg) | 3 months
  Pulse pressure (PP) is collected via home-based blood pressure measurement (HBPM) using a validated semi-automatic arm cuff device. HBPM will be performed according to the recommendations of the European Society of Hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Jauch-Chara, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No